CLINICAL TRIAL: NCT07301879
Title: Validation Study of the WB6Dim (Libellules) Digital Self-Assessment Tool for Well-Being Using Gold-Standard Psychometric Scales
Brief Title: Digital Self-Assessment of Well-Being: Validation of the Libellules Tool Against Gold-Standard Psychological Scales
Status: Completed | Type: Observational
Sponsor: Clover Link (Industry)
Responsible Party: Sponsor
Other Study IDs: WB6Dim
Record Dates: First submitted 2025-11-17; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Psychological Well Being
Keywords: Well-being, Self-assessment; Quality of life; Health promotion; Stress perception; Workplace well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A - Standard self-assessment: Participants complete the digital self-assessment "Libellules / WB6Dim" at baseline (T0) and after 14 days (T14) without any additional intervention. This group serves as the control for test-retest reliability and internal consistency analyses.
- Cohort B - Self-assessment + micro-intervention: Participants complete the same digital self-assessment "Libellules / WB6Dim" at baseline (T0) and after 14 days (T14), with a short preventive video intervention (guided breathing exercise). This group is used to explore the tool's sensitivity to change and short-term preventive impact.

SUMMARY:
The Libellules (WB6Dim) study aims to validate a digital self-assessment tool for measuring individual well-being across six dimensions: sleep and recovery, emotional climate, self-esteem, perceived autonomy, energy reservoir, and hyperconnection.

This observational study includes approximately 800 adult participants divided into two cohorts: one group completes the self-assessment tool only, while the other group additionally performs a brief video-based relaxation exercise during the 15-day interval between evaluations.

Each participant completes the Libellules questionnaire and a set of validated gold-standard psychometric scales (including PSS-10, ISI-7, CFQ, SAS-SV, and PIUQ-9) at baseline and after 15 days.

The primary objective is to evaluate the convergent validity, internal consistency, and test-retest reliability of the Libellules items compared with established instruments. The study is fully anonymous, non-interventional, and conducted in compliance with data protection regulations (CNIL, GDPR).

DETAILED DESCRIPTION:
Digital self-assessment tools are increasingly used in preventive health, workplace well-being programs, and population-level monitoring. However, most validated questionnaires currently available were designed for clinical or academic settings and rely on long item batteries that are difficult to deploy repeatedly in everyday contexts. The WB6Dim (Libellules) instrument was created to address this limitation by providing a brief, intuitive, and multidimensional representation of individual well-being suitable for large-scale, low-burden use.

The tool produces six numerical indicators-sleep and recovery, emotional climate, self-esteem, perceived autonomy, energy reservoir, and hyperconnection-derived from a short set of subjective items. During development, particular attention was given to clarity of wording, reduction of respondent fatigue, and the ability for individuals to understand and monitor their own "profile" over time. The instrument is fully digital and designed to be completed in under ten minutes, making it compatible with routine preventive practices.

The aim of the present study is to characterize the psychometric behavior of these digital indicators when used in real-life conditions. Because the tool is intended for repeated, short-interval use outside clinical contexts, the study examines how the indicators behave when measured twice over a two-week period. A two-cohort structure was employed to observe the natural stability of scores under standard conditions and to compare this with the evolution of scores in participants who voluntarily engaged with a brief relaxation video made available between the two time points. This simple stimulus was not intended as a clinical or therapeutic intervention but allowed exploration of short-term sensitivity while preserving the non-interventional nature of the study.

Data collection procedures were designed to guarantee complete anonymity. The platform was configured not to record IP addresses, names, emails, device identifiers, or free-text responses containing personal data. Only numerical questionnaire responses and non-identifying demographic categories were stored. This approach ensured compliance with GDPR and French CNIL requirements for anonymous observational research and removed the need for medical ethics board review.

The analytical approach focuses on commonly used psychometric properties relevant to short digital instruments. These include descriptive statistics, internal consistency of each dimension, temporal reproducibility between the two assessments, and correlations between the Libellules indicators and established psychometric scales covering conceptually related domains. All analyses were based exclusively on de-identified numerical data collected at baseline and follow-up. The purpose of these analyses is to document the measurement behavior of the six digital indicators and to determine whether their structure is compatible with future use in preventive, occupational, and public health contexts where rapid and repeated assessment is required.

The study does not involve clinical evaluation, diagnosis, treatment allocation, biological sampling, or medical follow-up. It provides foundational data for the future refinement of the WB6Dim instrument and for the development of scalable, user-friendly digital tools aimed at supporting well-being awareness and preventive initiatives at the individual and organizational level.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Able to read and understand French
* Access to an internet-connected device (computer, tablet, or smartphone)
* Willing to complete the digital self-assessment "Libellules / WB6Dim" at baseline and after 14 days
* Consent to anonymous data collection and analysis for research purposes

Exclusion Criteria:

* Individuals under 18 years of age
* Inability to read or understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult volunteers recruited from the general working population in France, including employees and independent workers participating in a health and well-being prevention program. Participants are not selected based on medical conditions but on their willingness to engage in a digital self-assessment of well-being. The cohort includes both men and women from diverse professional sectors, representing a broad spectrum of stress exposure, lifestyle, and occupational settings.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2025-10-09 (Actual); Primary Completion 2025-10-12 (Actual); Study Completion 2025-10-26 (Actual)

PRIMARY OUTCOMES:
Internal Consistency (Cronbach's Alpha) of the WB6Dim Sleep and Recovery dimension | From baseline (T0) to day 14 (T14).
  Evaluation of the internal consistency (Cronbach's alpha) of the Sleep and Recovery well-being dimension assessed by the Libellules / WB6Dim digital questionnaire.
  Score range: From 0 to 100. Interpretation: The higher the score, the stronger your resources. Higher scores reflect better balance.
Internal Consistency (Cronbach's Alpha) of the WB6Dim Emotional Climate dimension | From baseline (T0) to day 14 (T14).
  Evaluation of the internal consistency (Cronbach's alpha) of the Emotional Climate well-being dimension assessed by the Libellules / WB6Dim digital questionnaire.
  Score range: From 0 to 100. Interpretation: The higher the score, the stronger your resources. Higher scores reflect better balance.
Internal Consistency (Cronbach's Alpha) of the WB6Dim Energy Reservoir dimension | From baseline (T0) to day 14 (T14).
  Evaluation of the internal consistency (Cronbach's alpha) of the Energy Reservoir well-being dimension assessed by the Libellules / WB6Dim digital questionnaire.
  Score range: From 0 to 100. Interpretation: The higher the score, the stronger your resources. Higher scores reflect better balance.
Internal Consistency (Cronbach's Alpha) of the WB6Dim Perceived Autonomy dimension | From baseline (T0) to day 14 (T14).
  Evaluation of the internal consistency (Cronbach's alpha) of the Perceived Autonomy well-being dimension assessed by the Libellules / WB6Dim digital questionnaire.
  Score range: From 0 to 100. Interpretation: The higher the score, the stronger your resources. Higher scores reflect better balance.
Internal Consistency (Cronbach's Alpha) of the WB6Dim Self-Esteem dimension | From baseline (T0) to day 14 (T14).
  Evaluation of the internal consistency (Cronbach's alpha) of the Self-Esteem well-being dimension assessed by the Libellules / WB6Dim digital questionnaire.
  Score range: From 0 to 100. Interpretation: The higher the score, the stronger your resources. Higher scores reflect better balance.
Internal Consistency (Cronbach's Alpha) of the WB6Dim Internal Tension dimension | From baseline (T0) to day 14 (T14).
  Evaluation of the internal consistency (Cronbach's alpha) of the Internal Tension well-being dimension assessed by the Libellules / WB6Dim digital questionnaire.
  Score range: From 0 to 100. Interpretation: The higher the score, the stronger the tension. Lower scores reflect better balance.
Internal Consistency (Cronbach's Alpha) of the WB6Dim Hyperconnection dimension | From baseline (T0) to day 14 (T14).
  Evaluation of the internal consistency (Cronbach's alpha) of the Hyperconnection well-being dimension assessed by the Libellules / WB6Dim digital questionnaire.
  Score range: From 0 to 100. Interpretation: The higher the score, the stronger the hyperconnection. Lower scores reflect better balance.
Internal Consistency (Cronbach's Alpha) of the WB6Dim Cognitive Saturation dimension | From baseline (T0) to day 14 (T14).
  Evaluation of the internal consistency (Cronbach's alpha) of the Cognitive Saturation well-being dimension assessed by the Libellules / WB6Dim digital questionnaire.
  Score range: From 0 to 100. Interpretation: The higher the score, the stronger the saturation. Lower scores reflect better balance.
Test-Retest Reliability (Intraclass Correlation Coefficient) of the WB6Dim Sleep and Recovery dimension | Day 0 to Day 14
  Evaluation of the temporal stability of the Sleep and Recovery well-being dimension assessed by the Libellules / WB6Dim digital questionnaire over a 14-day interval.
  Score range: Intraclass Correlation Coefficient (ICC), from 0 to 1. Interpretation: Higher ICC values indicate greater temporal stability of the score over time.
Test-Retest Reliability (Intraclass Correlation Coefficient) of the WB6Dim Self-Esteem dimension | Day 0 to Day 14.
  Evaluation of the temporal stability of the Self-Esteem well-being dimension assessed by the Libellules / WB6Dim digital questionnaire over a 14-day interval.
  Score range: Intraclass Correlation Coefficient (ICC), from 0 to 1. Interpretation: Higher ICC values indicate greater temporal stability of the score over time.
Test-Retest Reliability (Intraclass Correlation Coefficient) of the WB6Dim Perceived Autonomy dimension | Day 0 to Day 14.
  Evaluation of the temporal stability of the Perceived Autonomy well-being dimension assessed by the Libellules / WB6Dim digital questionnaire over a 14-day interval.
  Score range: Intraclass Correlation Coefficient (ICC), from 0 to 1. Interpretation: Higher ICC values indicate greater temporal stability of the score over time.
Test-Retest Reliability (Intraclass Correlation Coefficient) of the WB6Dim Energy Reservoir dimension | Day 0 to Day 14.
  Evaluation of the temporal stability of the Energy Reservoir well-being dimension assessed by the Libellules / WB6Dim digital questionnaire over a 14-day interval.
  Score range: Intraclass Correlation Coefficient (ICC), from 0 to 1. Interpretation: Higher ICC values indicate greater temporal stability of the score over time.
Test-Retest Reliability (Intraclass Correlation Coefficient) of the WB6Dim Internal Tension dimension | Day 0 to Day 14.
  Evaluation of the temporal stability of the Internal Tension well-being dimension assessed by the Libellules / WB6Dim digital questionnaire over a 14-day interval.
  Score range: Intraclass Correlation Coefficient (ICC), from 0 to 1. Interpretation: Higher ICC values indicate greater temporal stability of the score over time.
Test-Retest Reliability (Intraclass Correlation Coefficient) of the WB6Dim Hyperconnection dimension | Day 0 to Day 14.
  Evaluation of the temporal stability of the Hyperconnection well-being dimension assessed by the Libellules / WB6Dim digital questionnaire over a 14-day interval.
  Score range: Intraclass Correlation Coefficient (ICC), from 0 to 1. Interpretation: Higher ICC values indicate greater temporal stability of the score over time.
Test-Retest Reliability (Intraclass Correlation Coefficient) of the WB6Dim Cognitive Saturation dimension | Day 0 to Day 14.
  Evaluation of the temporal stability of the Cognitive Saturation well-being dimension assessed by the Libellules / WB6Dim digital questionnaire over a 14-day interval.
  Score range: Intraclass Correlation Coefficient (ICC), from 0 to 1. Interpretation: Higher ICC values indicate greater temporal stability of the score over time.

SECONDARY OUTCOMES:
Convergent Validity of the WB6Dim Sleep and Recovery dimension vs Insomnia Severity Index (ISI-7) | Day 0 and Day 14
  Outcome Measure:
  Correlation coefficient between the WB6Dim Sleep and Recovery dimension score and the Insomnia Severity Index (ISI-7) score.
  Description:
  Assessment of convergent validity through correlation analysis between the Sleep and Recovery dimension of the Libellules / WB6Dim digital questionnaire and insomnia severity as measured by the Insomnia Severity Index (ISI-7).
  Higher scores on the Sleep and Recovery dimension are expected to be associated with lower ISI-7 scores, reflecting better sleep quality and recovery.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Sleep and Recovery dimension vs Perceived Stress Scale (PSS-10) | Day 0 and Day 14.
  Outcome Measure:
  Correlation coefficient between the WB6Dim Sleep and Recovery dimension score and the Perceived Stress Scale (PSS-10) score.
  Description:
  Assessment of convergent validity through correlation analysis between the Sleep and Recovery dimension of the Libellules / WB6Dim digital questionnaire and perceived stress as measured by the PSS-10.
  Higher scores on the Sleep and Recovery dimension are expected to be associated with lower perceived stress levels.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Sleep and Recovery dimension vs WHO-5 Well-Being Index | Day 0 and Day 14.
  Outcome Measure:
  Correlation coefficient between the WB6Dim Sleep and Recovery dimension score and the WHO-5 Well-Being Index score.
  Description:
  Assessment of convergent validity through correlation analysis between the Sleep and Recovery dimension of the Libellules / WB6Dim digital questionnaire and general well-being as measured by the WHO-5 Well-Being Index.
  Higher scores on the Sleep and Recovery dimension are expected to be associated with higher WHO-5 well-being scores.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Self-Esteem dimension vs Rosenberg Self-Esteem Scale (RSES) | Day 0 and Day 14.
  Outcome Measure:
  Correlation coefficient between the WB6Dim Self-Esteem dimension score and the Rosenberg Self-Esteem Scale (RSES) score.
  Description:
  Assessment of convergent validity through correlation analysis between the Self-Esteem dimension of the Libellules / WB6Dim digital questionnaire and self-esteem as measured by the RSES.
  Higher scores on the Self-Esteem dimension are expected to be associated with higher self-esteem levels.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Self-Esteem dimension vs WHO-5 Well-Being Index | Day 0 and Day 14.
  Outcome Measure:
  Correlation coefficient between the WB6Dim Self-Esteem dimension score and the WHO-5 Well-Being Index score.
  Description:
  Assessment of convergent validity through correlation analysis between the Self-Esteem dimension of the Libellules / WB6Dim digital questionnaire and general psychological well-being as measured by the WHO-5 Well-Being Index.
  Higher scores on the Self-Esteem dimension are expected to be associated with higher WHO-5 well-being scores.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Perceived Autonomy dimension vs Basic Psychological Needs Satisfaction (BPNS) | Day 0 and Day 14.
  Outcome Measure:
  Correlation coefficient between the WB6Dim Perceived Autonomy dimension score and the autonomy-related subscale of the Basic Psychological Needs Satisfaction (BPNS) scale.
  Description:
  Assessment of convergent validity through correlation analysis between the Perceived Autonomy dimension of the Libellules / WB6Dim digital questionnaire and psychological needs satisfaction as measured by the BPNS scale.
  Higher scores on the Perceived Autonomy dimension are expected to be associated with higher satisfaction of psychological autonomy needs.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Energy Reservoir dimension vs WHO-5 Well-Being Index | Day 0 and Day 14.
  Outcome Measure:
  Correlation coefficient between the WB6Dim Energy Reservoir dimension score and the WHO-5 Well-Being Index score.
  Description:
  Assessment of convergent validity through correlation analysis between the Energy Reservoir dimension of the Libellules / WB6Dim digital questionnaire and general well-being as measured by the WHO-5 Well-Being Index.
  Higher scores on the Energy Reservoir dimension are expected to be associated with higher well-being levels.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Energy Reservoir dimension vs Copenhagen Burnout Inventory (CBI) | Day 0 and Day 14
  Outcome Measure:
  Correlation coefficient between the WB6Dim Energy Reservoir dimension score and the Personal Burnout subscale of the Copenhagen Burnout Inventory (CBI).
  Description:
  Assessment of convergent validity through correlation analysis between the Energy Reservoir dimension of the Libellules / WB6Dim digital questionnaire and burnout-related exhaustion as measured by the CBI Personal Burnout subscale.
  Higher scores on the Energy Reservoir dimension are expected to be associated with lower burnout scores.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Internal Tension dimension vs Perceived Stress Scale (PSS-10) | Day 0 and Day 14
  Outcome Measure:
  Correlation coefficient between the WB6Dim Internal Tension dimension score and the Perceived Stress Scale (PSS-10) score.
  Description:
  Assessment of convergent validity through correlation analysis between the Internal Tension dimension of the Libellules / WB6Dim digital questionnaire and perceived stress.
  Higher scores on the Internal Tension dimension are expected to be associated with higher perceived stress levels.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Internal Tension dimension vs Copenhagen Burnout Inventory (CBI) | Day 0 and Day 14
  Outcome Measure:
  Correlation coefficient between the WB6Dim Internal Tension dimension score and the Copenhagen Burnout Inventory (CBI) Personal and Work Burnout subscales.
  Description:
  Assessment of convergent validity through correlation analysis between the Internal Tension dimension of the Libellules / WB6Dim digital questionnaire and burnout-related strain.
  Higher scores on the Internal Tension dimension are expected to be associated with higher burnout scores.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Internal Tension dimension vs UCLA Loneliness Scale (UCLA-3) | Day 0 and Day 14
  Outcome Measure:
  Correlation coefficient between the WB6Dim Internal Tension dimension score and the UCLA Loneliness Scale (UCLA-3) score.
  Description:
  Assessment of convergent validity through correlation analysis between the Internal Tension dimension of the Libellules / WB6Dim digital questionnaire and perceived loneliness.
  Higher scores on the Internal Tension dimension are expected to be associated with higher loneliness scores.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Hyperconnection dimension vs Smartphone Addiction Scale - Short Version (SAS-SV) | Day 0 and Day 14
  Outcome Measure:
  Correlation coefficient between the WB6Dim Hyperconnection dimension score and the Smartphone Addiction Scale - Short Version (SAS-SV) score.
  Description:
  Assessment of convergent validity through correlation analysis between the Hyperconnection dimension of the Libellules / WB6Dim digital questionnaire and problematic smartphone use.
  Higher scores on the Hyperconnection dimension are expected to be associated with higher levels of problematic smartphone use.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Hyperconnection dimension vs Cognitive Failures Questionnaire (CFQ-9) | Day 0 and Day 14
  Outcome Measure:
  Correlation coefficient between the WB6Dim Hyperconnection dimension score and the Cognitive Failures Questionnaire - short form (CFQ-9) score.
  Description:
  Assessment of convergent validity through correlation analysis between the Hyperconnection dimension of the Libellules / WB6Dim digital questionnaire and cognitive difficulties.
  Higher scores on the Hyperconnection dimension are expected to be associated with higher cognitive failure scores.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Cognitive Saturation dimension vs Cognitive Failures Questionnaire (CFQ-9) | Day 0 and Day 14
  Outcome Measure:
  Correlation coefficient between the WB6Dim Cognitive Saturation dimension score and the Cognitive Failures Questionnaire - short form (CFQ-9) score.
  Description:
  Assessment of convergent validity through correlation analysis between the Cognitive Saturation dimension of the Libellules / WB6Dim digital questionnaire and cognitive overload and attentional difficulties.
  Higher scores on the Cognitive Saturation dimension are expected to be associated with higher cognitive failure scores.
  Measure Type: Correlation coefficient (r)
Convergent Validity of the WB6Dim Cognitive Saturation dimension vs Perceived Stress Scale (PSS-10) | Day 0 and Day 14
  Outcome Measure:
  Correlation coefficient between the WB6Dim Cognitive Saturation dimension score and the Perceived Stress Scale (PSS-10) score.
  Description:
  Assessment of convergent validity through correlation analysis between the Cognitive Saturation dimension of the Libellules / WB6Dim digital questionnaire and perceived stress.
  Higher scores on the Cognitive Saturation dimension are expected to be associated with higher perceived stress levels.
  Measure Type: Correlation coefficient (r)

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique RETORNAZ, MD, PhD, Study Chair — European Hospital, Unit of Care and Research in Internal Medicine and Infectious Diseases.
Locations (1):
- Clover Link, Bandol, France

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because all collected data are fully anonymized and aggregated for psychometric and statistical analyses only. No identifiable personal data are stored